CLINICAL TRIAL: NCT00371488
Title: Phase I Study of Lapatinib in Combination With Trastuzumab
Brief Title: GW572016 Combined With Trastuzumab For The Treatment Of Previously Trastuzumab-Treated Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF105635
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms, Breast
Keywords: ErbB2; Stage IV breast cancer; ErbB1; breast cancer; lapatinib; Herceptin; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GW572016 in combination with trastuzumab (Experimental): Lapatinib:
  A specified dose of lapatinib will be orally taken once daily, at least one hour before or one hour after the morning meal. Lapatinib should be taken at the same time of day wherever possible.
  The starting dose of lapatinib should be 750 mg/day, which will be increased to 1000 mg/day (dose escalation group) according to the dose escalation criteria.
  Trastuzumab:
  Trastuzumab (4 mg/kg/day in the first week and 2 mg/kg/day for the 2nd and subsequent weeks) will be administered by intravenous infusion over at least 90 minutes immediately after administration of lapatinib. The fifth (Day 36) and subsequent doses may be administered up to 3 days after the scheduled date. In this case, however, the all following doses should be administered at one-week intervals.
  Interventions: Drug: GW572016 oral tablets

INTERVENTIONS:
Drug: GW572016 oral tablets — Tablets contain 405mg of lapatinib ditosylate monohydrate, equivalent to 250mg lapatinib free base per tablet. Oval, orange, film-coated tablets.

SUMMARY:
This is two-part study (Phase I/Phase II). Part I is designed to find the optimal (best) doses of GW572016 and trastuzumab when given together,Part II is designed to evaluate the tumor response rate (shrinkage or lack of growth) in patients receiving lapatinib and trastuzumab.

ELIGIBILITY:
Inclusion criteria:

* Patients with confirmed breast cancer who have received prior trastuzumab.
* Patients must have adequate blood, liver, and kidney function and either be fully active or restricted only in performing strenuous activity.
* Female patients of child-bearing potential must be willing to abstain from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication or be willing to consistently and correctly use an acceptable method of birth control.

Exclusion criteria:

* Patients with certain heart problems.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-04-06 (Actual); Primary Completion 2007-12-10 (Actual); Study Completion 2007-12-10 (Actual)

PRIMARY OUTCOMES:
Optimal doses and toleration of the two drugs administered together Tumor progression measured by radiological imaging 4-8 weekly | 6 Months
  To confirm the safety and tolerability of the recommended dose of lapatinib in combination with trastuzumab which was determined in a preceding overseas study, and to determine the recommended dose in Japan.

SECONDARY OUTCOMES:
Clinical benefit Time to tumor response Length of response Time to progression of cancer 6 month progression free survival Overall survival as well as specific biomarkers in tumor tissue | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

REFERENCES:
- See also: Results for study EGF105635 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/EGF105635?search=study&search_terms=EGF105635#rs